CLINICAL TRIAL: NCT04472728
Title: Adaptive Design Phase 2 to 3, Randomized, Double-blind, to Evaluate Safety, Efficacy, Pharmacokinetics and Pharmacodynamics of BIO101 in the Prevention of the Respiratory Deterioration in Hospitalized COVID-19 Patients
Brief Title: Testing the Efficacy and Safety of BIO101 for the Prevention of Respiratory Deterioration in COVID-19 Patients
Acronym: COVA
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lack of eligible patients due to lower number of Covid-19 cases in all involved sites.
Sponsor: Biophytis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIO101-CL05
Record Dates: First submitted 2020-07-06; First posted 2020-07-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2022-04

CONDITIONS: Covid-19; SARS-CoV2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BIO101 (Experimental): BIO101 350 mg bid
  Interventions: Drug: BIO101
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIO101 — BIO101 capsules
  Other Names: Sarconeos (BIO101)
  Arms: BIO101
Drug: Placebo — placebo capsules
  Other Names: Sarconeos (placebo)
  Arms: Placebo

SUMMARY:
The COVA clinical study is a global multicentric, double-blind, placebo-controlled, group sequential and adaptive 2 parts phase 2-3 study targeting in patients with SARS-CoV-2 pneumonia. Part 1 is a Phase 2 exploratory Proof of Concept (PoC) study to provide preliminary data on the activity, safety and tolerability of BIO101 in the target population. Part 2 is a phase 3 pivotal randomized study to provide further evidence of safety and efficacy of BIO101 after 28 days of double-blind dosing. BIO101 is the investigational new drug that activates the Mas receptor (MasR) through the protective arm of the Renin Angiotensin System (RAS).

DETAILED DESCRIPTION:
Biophytis is developing BIO101, an investigational new drug, an oral preparation of immediate-release 20-hydroxyecdysone (20E) at ≥ 97% purity. BIO101 activates MasR on the protective arm of the Renin Angiotensin System (RAS). The engagement of MasR by BIO101 is responsible for a number of preclinical beneficial activities in normal and pathological contexts.

The COVA clinical study is a global, multicentric, double-blind, placebo-controlled, group sequential and adaptive 2 parts phase 2-3 study in participants with SARS-CoV-2 pneumonia. Part 1 is a Phase 2 exploratory Proof of Concept (PoC) study to provide preliminary data on the activity, safety and tolerability of BIO101 in the target population. Part 2 is a phase 3 pivotal randomized study to provide further evidence of safety and efficacy of BIO101 after 28 days of dosing.

The trial will use an adaptive design based on pre-specified criteria, using an independent external Data Monitoring Committee (DMC) to monitor safety, efficacy, and review data at appropriate intervals to allow the initiation of the confirmatory part of the study.

The general objectives of the study are:

* The purpose of Part 1 is to obtain preliminary indication of activity of BIO101, in preventing respiratory deterioration in the target population (50 patients, age ≥ 55 years) and provide preliminary data on the safety and tolerability of BIO101 in the target population
* The purpose of Part 2 is to re-assess the sample size that is needed for the confirmatory part of the study and to provide confirmation on the benefit of BIO101 and safety in the larger target population (up to 310 patients)

ELIGIBILITY:
Inclusion Criteria:

1. Age: 45 and older (in France: 55 and older)
2. A confirmed diagnosis of COVID-19 infection, within the last 28 days, prior to randomization, as determined by PCR or other approved commercial or public health assay, in a specimen as specified by the test used.
3. Hospitalized, in observation or planned to be hospitalized due to COVID-19 infection symptoms with anticipated hospitalization duration >=3 days

   a. Patients can be included even if treated with: oxygen supplementation, High-flow oxygen (HFO2), BiPAP and CPAP
4. With evidence of pneumonia based on all of the following:

   1. Clinical findings on a physical examination
   2. Respiratory symptoms developed within the past 14 days
5. With evidence of respiratory decompensation that started not more than 7 days before start of study medication and present at screening, meeting one of the following criteria, as assessed by healthcare staff:

   1. Tachypnea: ≥25 breaths per minute
   2. Arterial oxygen saturation ≤92%
   3. A special note should be made if there is suspicion of COVID-19- related myocarditis or pericarditis, as the presence of these is a stratification criterion
6. Without a significant deterioration in liver function tests:

   1. ALT and AST ≤ 5x upper limit of normal (ULN)
   2. Gamma-glutamyl transferase (GGT) ≤ 5x ULN
   3. Total bilirubin ≤ 5×ULN
7. Willing to participate and able to sign an informed consent form (ICF)
8. Female subjects should be:

   at least 5 years post-menopausal (i.e., persistent amenorrhea 5 years in the absence of an alternative medical cause) or surgically sterile; OR
   1. Have a negative urine pregnancy test at screening
   2. Be willing to use a contraceptive method as outlined in inclusion criterion 9 from screening to 30 days after last dose.
9. Male subjects who are sexually active with a female partner must agree to the use of an effective method of birth control throughout the study and until 3 months after the last administration of investigational product; Note: medically acceptable methods of contraception that may be used by the subject and/or partner include combined oral contraceptive, contraceptive vaginal ring, contraceptive injection, intrauterine device, etonogestrel implant, each supplemented with a condom, as well as sterilization and vasectomy.
10. Male subjects must agree not to donate sperm for the purpose of reproduction throughout the study and until 3 months after the last administration of investigational product;
11. For France only: Being affiliated with a European Social Security.

Exclusion Criteria:

1. Not needing or not willing to remain in a healthcare facility during the entire study medication (i.e. while receiving study medication)
2. Moribund condition (death likely in days) or not expected to survive for >7 days - due to other and non-COVID-19 related conditions
3. Patient on invasive mechanical ventilation via an endotracheal tube, or extracorporeal membrane oxygenation (ECMO)
4. Patient within 7 days of participating in other therapeutic clinical trial with angiotensin-converting-enzyme inhibitors (ACEi), angiotensin receptor blockers (ARB) or recombinant ACE-2
5. Patient not able to take medications by mouth (as capsules or as a powder, mixed in water).
6. Disallowed concomitant medication:

   a. Consumption of any herbal products containing 20-hydroxyecdysone and derived from Leuzea carthamoides; Cyanotis vaga or Cyanotis arachnoidea is not allowed (e.g. performance enhancing agents)
7. Any known hypersensitivity to any of the ingredients, or excipients of the study medication, BIO101
8. In France:

   * Non-affiliation to compulsory French social security scheme (beneficiary or right-holder)
   * Being under tutelage or legal guardianship

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
End-of-Part 1 interim analysis: Proportion of subjects with all cause mortality or with respiratory failure. | up to 28 days
  For interim analysis intended to obtain indication of activity of BIO101.
  Primary endpoint:
  • Proportion of subjects with negative events, of either of the following:
  * All-cause mortality
  * Respiratory failure, defined as any of the following:
  Requiring mechanical ventilation (including cases that will not be intubated due to resource restrictions and triage) Requiring ECMO
For part-2 sample size interim analysis: Proportion of subjects with all cause mortality or with respiratory failure. | up to 28 days
  For sample size re-assessment for part 2, time frame - up to 28 days:
  • Proportion of participants with negative events, of either of the following:
  * All-cause mortality
  * Respiratory failure, defined as any of the following:
  Requiring mechanical ventilation (including cases that will not be intubated due to resource restrictions and triage) Requiring ECMO
For the final analysis: Proportion of subjects with all cause mortality or respiratory failure. | up to 28 days
  • Proportion of participants with of subjects with negative events, of either of the following.
  * All-cause mortality
  * Respiratory failure, defined as any of the following:
  Mechanical ventilation (including cases that will not be intubated due to resource restrictions and triage) Requiring ECMO

SECONDARY OUTCOMES:
Interim analysis; indication of activity of BIO101: Oxygen saturation by pulse oximetry (SpO2) SpO2 / Fraction of inspired oxygen (FiO2) ratio | 28 days
  • SpO2/FiO2
Interim analysis; indication of activity of BIO101: Inflammatory markers | 28 days
  • Inflammatory markers including:
  * IL 6
  * TNFα
  * D-dimer
Interim analysis; indication of activity of BIO101: Renin Angiotensin System biomarkers | 28 days
  • Renin Angiotensin System biomarkers:
  * Angiotensin 2
  * Angiotensin-converting enzyme (ACE) levels
Key secondary endpoint for final analysis: Proportion of participants with positive events | Up to 28 days
  • official discharge from hospital care by the department due to improvement in participant condition (self-discharge by participant is not considered a positive event)
Additional secondary endpoints for final analysis: Respiratory function | 28 days
  Oxygen saturation in arterial blood, measured by pulse-oximetry (SpO2) SpO2/FiO2 Proportion of participants with CPAP/BiPAP events, defined as requiring CPAP/BiPAP/HFO2 in participants entering the study on low flow oxygen)
Additional secondary endpoints for final analysis:proportion of patients who experienced negative events | 28 days
  Time to events, of either of the following:
  * All-cause mortality
  * Respiratory failure, defined as any of the following: Requiring mechanical ventilation (including cases that will not be intubated due to resource restrictions and triage); Requiring ECMO; • Proportion of participants with CPAP/BiPAP/HFO2 events, defined as requiring CPAP/BiPAP/HFO2 in participants entering the study on low flow oxygen)
Additional secondary endpoint for final analysis: The National Early Warning Score 2 (NewS2): | 28 days
  National Early Warning Score 2 (NewS2): scores: 0-7
Additional secondary endpoint for final analysis: Population Pharmacokinetics study (pop-PK) | 1day
  Cmax: Peak Plasma concentration
Additional secondary endpoint : Population Pharmacokinetics study (pop-PK) | 1 day
  tmax: Time to reach peak plasma concentration
Additional secondary endpoint: Population Pharmacokinetics study (pop-PK) | 1 day
  AUC: Area under the plasma concentration versus time curve
Additional secondary endpoint: Proportion of participants with events of all-cause mortality | Up to 28 days
  Proportion of participants with events of all-cause mortality
Additional secondary endpoint: time to event: negative events | Up to 28 days
  Time to events, of either of the following:
  * All-cause mortality
  * Respiratory failure, defined as any of the following:
    * Requiring mechanical ventilation (including cases that will not be intubated due to resource restrictions and triage)
    * Requiring ECMO
Additional secondary endpoint: time to event: positive events | Up to 28 days
  Time to event: official discharge from hospital care due to improvement

CONTACTS AND LOCATIONS:
Overall Officials: Capucine Morelot-Panzini, MD, Principal Investigator — Département R3S GHU APHP-Sorbonne Université, Pitié Salpetrière
Locations (22):
- United States (6):
  - Abrazo Health, Phoenix, Arizona
  - University of California, Irvine, Irvine, California
  - Barnum Medical Research, Inc. 1029 Keyser Ave Suite H, Natchitoches, Louisiana
  - Beaumont Health, Royal Oak, Michigan
  - United Health Services Hospitals, Johnson City, New York
  - WellSpan Health, York, Pennsylvania
- Belgium (3):
  - CHU Saint-Pierre, Brussels
  - AZ-Sint Maarten, Mechelen
  - CHU CLU Namur (Saint-Elisabeth) Place Louise Godin, Namur
- Brazil (6):
  - Hospital Vera Cruz, Belo Horizonte, Minas Gerais
  - Santa Casa de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Municipal de Barueri Dr. Francisco Moran, Barueri, São Paulo
  - Hospital e Maternidade Celso Pierro - PUCCAMP, Campinas, São Paulo
  - Hospital de Base Da Faculdade de Medicina de São José Do Rio Preto, São José do Rio Preto, São Paulo
  - Avenida Dr. Enéas de Carvalho Aguiar, 44 - Centro de Pesquisa Clínica Prof. Dr. Fúlvio Pileggi - Bloco 1 - 1º Andar, São Paulo
- France (6):
  - Unité ambulatoire Service de Pneumologie, Médecine Intensive et Réanimation (SPMIR) 47-83 Boulevard de l'Hôpital, Paris, Paris Cedex 13
  - Centre Hospitalier Argenteuil, Argenteuil
  - Centre Hospitalier Universitaire Bordeaux, Bordeaux
  - Centre Hospitalier Rene Dubos, Cergy-Pontoise
  - Centre Hospitalier Départemental de Vendée, La Roche-sur-Yon
  - Hôpital Pitié-Salpêtrière, 47 bd de l'Hôpital, 75013 Paris, Paris
- FDI Clinical Research - San Juan City Hospital, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lobo SM, Plantefeve G, Nair G, Joaquim Cavalcante A, Franzin de Moraes N, Nunes E, Barnum O, Berdun Stadnik CM, Lima MP, Lins M, Hajjar LA, Lipinski C, Islam S, Ramos F, Simon T, Martinot JB, Guimard T, Desclaux A, Lioger B, Neuenschwander FC, DeSouza Paolino B, Amin A, Acosta SA, Dilling DF, Cartagena E, Snyder B, Devaud E, Barreto Berselli Marinho AK, Tanni S, Milhomem Beato PM, De Wit S, Selvan V, Gray J, Fernandez R, Pourcher V, Maddox L, Kay R, Azbekyan A, Chabane M, Tourette C, Esmeraldino LE, Dilda PJ, Lafont R, Mariani J, Camelo S, Rabut S, Agus S, Veillet S, Dioh W, van Maanen R, Morelot-Panzini C. Efficacy of oral 20-hydroxyecdysone (BIO101), a MAS receptor activator, in adults with severe COVID-19 (COVA): a randomized, placebo-controlled, phase 2/3 trial. EClinicalMedicine. 2024 Jan 3;68:102383. doi: 10.1016/j.eclinm.2023.102383. eCollection 2024 Feb. PMID 38545090
- [Derived] Dioh W, Chabane M, Tourette C, Azbekyan A, Morelot-Panzini C, Hajjar LA, Lins M, Nair GB, Whitehouse T, Mariani J, Latil M, Camelo S, Lafont R, Dilda PJ, Veillet S, Agus S. Testing the efficacy and safety of BIO101, for the prevention of respiratory deterioration, in patients with COVID-19 pneumonia (COVA study): a structured summary of a study protocol for a randomised controlled trial. Trials. 2021 Jan 11;22(1):42. doi: 10.1186/s13063-020-04998-5. PMID 33430924